CLINICAL TRIAL: NCT06871176
Title: [68Ga]Ga-PentixaFor (CXCR4) PET/MR for Initial Staging and Follow up in Multiple Myeloma: Prospective Comparison With Standard of Care PET/CT and Evaluation of Therapy Influence
Brief Title: PET/MR Scan With [68Ga]Ga-PentixaFor (CXCR4) vs Standard of Care (SOC) for Initial Staging and Follow up in Multiple Myeloma (MM)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-5828
Record Dates: First submitted 2025-02-27; First posted 2025-03-11 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, controlled, comparative study. Participants with newly diagnosed multiple myeloma will undergo both standard imaging (18F-FDG-PET/CT and MRI) and the investigational [68Ga]Ga-PentixaFor (CXCR4) PET/MR imaging. The study will assess the diagnostic accuracy and potential therapeutic influence of the CXCR4 PET/MR scan in comparison to the standard of care. The study will include both initial staging and follow-up imaging assessments, with an emphasis on how the new imaging modality influences treatment decisions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CXCR4-targeted [68Ga]Ga-PentixaFor PET/MR Imaging (Experimental): This arm involves patients undergoing the investigational imaging modality, CXCR4-targeted [68Ga]Ga-PentixaFor PET/MR, to evaluate its diagnostic, prognostic, and therapeutic value in comparison to standard imaging methods.
  Interventions: Drug: [68Ga]Ga-PentixaFor

INTERVENTIONS:
Drug: [68Ga]Ga-PentixaFor — [68Ga]Ga-PentixaFor will be administered intravenously using the recommended activity for adults which is up to 150 MBq (4 mCi) fixed dose. There is no weight adaption recommended in the literature.
  Other Names: CXCR4

SUMMARY:
Multiple myeloma is a disease mainly located in participants bones. Usually a participants physician arrives at this diagnosis by doing blood tests and ordering standard of care imaging tests (18F-FDG PET/CT and maybe additional MRI) to see how many bones (and/or other organs) are affected. While these two imaging tests are already very good, recent research indicates that even more precise imaging methods could be used to diagnose participants disease more precisely.

The purpose of this study is to learn if a combined PET/MR scan with a new radiotracer, [68Ga]Ga-PentixaFor, can provide more accurate and precise diagnostic information in patients with Multiple Myeloma, a type of cancer primarily affecting the bones.

This study aims to improve the accuracy of diagnosing and monitoring Multiple Myeloma using more advanced imaging techniques.

DETAILED DESCRIPTION:
The investigators will be focusing on Multiple Myeloma patients, a disease mainly located in the participants bones. The goal of this clinical trial is to evaluate the diagnostic and prognostic value of CXCR4-targeted PET/MR imaging in patients with Multiple Myeloma (MM), comparing it to the standard 18F-FDG-PET/CT and MRI imaging for the initial staging, follow-up, and treatment decision-making. The study will focus on newly diagnosed MM patients and those who may undergo stem cell transplantation.

The investigators will compare the performance of [68Ga]Ga-PentixaFor PET/MR to standard imaging methods (18F-FDG-PET/CT and MRI) to see if CXCR4-targeted imaging offers improved accuracy, better tumor detection, and a greater influence on treatment decisions.

This study aims to establish whether combining CXCR4-targeted PET/MR imaging could become a comprehensive diagnostic tool for MM, enhancing disease monitoring, guiding therapeutic decisions, and reducing patient burden by eliminating the need for multiple imaging sessions.

ELIGIBILITY:
Inclusion criteria

* Patient older than 18 years of age
* Clinical diagnosis of (nonsecretory, oligosecretory, suspicion for extramedullary MM) MM. MM diagnosis is based on IMWG (International Myeloma Working Group) criteria.No treatment received beyond first course of

Exclusion criteria

* Any contra-indications for MRI or 18F-FDG PET/CT imaging according to institutional guideline
* Pregnancy (will be ruled out as per institutional protocol)
* Inability to lie still in prone position in MRI for at least 30 min or PET/CT for at least 30 min
* Patients or unwilling to use contraception during study and breastfeeding women can also not partake in this study
* Inability to provide consent
* Any hypersensitivity or known allergy to any component of the investigational product ([68Ga]Ga-PentixaFor)No concomitant other malignant hemato-oncological disease being diagnosed (i.e. additional lymphoma or leukemia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2028-03-04 (Estimated); Study Completion 2028-03-04 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of CXCR4-targeted [68Ga]Ga-PentixaFor PET/MR Imaging Compared to Standard of Care Imaging | Baseline (at initial staging)
  This primary outcome will assess the diagnostic accuracy of the CXCR4-targeted [68Ga]Ga-PentixaFor PET/MR imaging in comparison to the standard 18F-FDG PET/CT and MRI imaging in newly diagnosed multiple myeloma (MM) patients. Specifically, the focus will be on the number of bone marrow myeloma manifestations detected by CXCR4 PET/MR compared to standard imaging, as well as the number of extra-osseous myeloma manifestations detected.

SECONDARY OUTCOMES:
Evaluating the Role of CXCR4-targeted Imaging in Treatment Decision Making Using a Questionnaire | Post-initial staging (before starting treatment)
  Using a questionnaire, the investigators aim to evaluate how hematologists make treatment decisions based on the addition of CXCR4 PET/MR imaging influences in MM patients, including adjustments in preconditioning, evaluation for radiotherapy, decisions for or against stem cell transplantation, and changes in follow-up schedules.
Evaluating the Role of CXCR4-targeted Imaging in Response Assessment Using a Questionnaire | 3 months after start of participants therapy for MM
  Using a questionnaire, the investigators aim to evaluate how hematologist assess how the availability of CXCR4 PET/MR affects decisions during therapy response assessment. This could include changes in imaging follow-up, supportive therapy decisions, or additional evaluations.
Gather data to inform on patient selection for theranostics studies | Baseline (initial staging)
  The investigators will collect all data measurements on imaging and disease characteristics from CXCR4 imaging and standard-of-care imaging, integrating these findings to form a comprehensive assessment of whether patients may be suitable candidates for theranostic studies
Monitoring for Adverse Events Related to Radiopharmaceutical Administration | 6 months (from baseline to final follow-up)
  Document any adverse events following the administration of the radiopharmaceutical [68Ga]Ga-PentixaFor during PET/MR imaging, including any potential side effects or safety concerns.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Veit-Haibach, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada